CLINICAL TRIAL: NCT06762028
Title: Exploring the Relationship Between L-dopa Responsiveness and Small Intestinal Microbiome in Parkinson's Disease
Acronym: LENSER
Status: Not yet recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: UCalgaryREB24-1779; POP24-11461 (Other Grant/Funding Number: Weston Family Foundation)
Record Dates: First submitted 2024-12-20; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: SIMBA; small intestine; L-dopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: SIMBA capsule — The small intestine microbiome aspiration (SIMBA) system is a single-use, ingestible passive capsule that allows for the non-invasive sampling of small intestinal contents. It is designed to open and adsorb intestinal content after having passed the acid stomach environment and to close mechanically before passing into the large bowel. It has distinct markers built in to allow radiographic tracking of its passage throughout the GI system.

SUMMARY:
The investigators hypothesize that small intestinal (SI) microbiome biomarkers predict the responsiveness to oral levodopa/carbidopa in people with Parkinson's disease (PwPD). The investigators will analyze the bacterial species and function of bacterial pathways influencing the responsiveness of PwPD to oral L-dopa. The investigators will pursue this goal using a reliable capsule system (SIMBA capsule, Nimble Science, Calgary, AB) that suitably captures SI luminal fluid for multi-omics analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 50-85 years old at time of on-site visit. (ages 81-85 will be assessed on a per case basis by the principal investigator)
2. Signed Informed consent.
3. Willing & able to comply with study procedures (including SIMBA capsule ingestion) and have study assessments performed.
4. Able to swallow a size-00 capsule (25mm length) in OFF state.
5. Diagnosis of idiopathic PD (Clinically Probable PD), including documented levodopa responsiveness.
6. Treatment with an immediate release levodopa formulation during the day at a stable dose for at least 2 months prior to enrollment.

Exclusion Criteria:

1. Any risk of capsule non-excretion related to intercurrent gastrointestinal conditions.
2. Use of any medications in the week prior to the on-site study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function.
3. History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration, e.g., SDQ score > 4.
4. Any concomitant or previous treatment (<2 months from on-site study visit) with significant anti-inflammatory or immune suppressant medication, e.g., DMARDs, biologicals or systemic corticosteroids, except non-chronic PRN use of an NSAID and/or 5-ASA (mesalazine) treatment.
5. Active cancer within 5 years.
6. Clinically significant immune deficiency (according to Investigator's judgement).
7. Antibiotic use (except for local use), ≤12 weeks prior to on-site study visit, or Fecal Microbiota Transplantation anytime in medical history.
8. Use of prebiotics, or probiotics ≤2 weeks prior to the on-site study visit.
9. Dementia in medical history.
10. Insulin-dependent diabetes mellitus.
11. Current Psychosis episode by clinical judgement based on anamnesis.
12. Pregnancy.
13. Alcohol or drug abuse.
14. Deep brain stimulation or Duodopa/Lecigon treatment.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with Parkinson disease fulfilling section criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of Part 3 score of the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) on L-dopa challenge test | Same day of study visit
  The primary outcome is the acute responsiveness to an immediate release L-dopa/carbidopa or L-dopa/benserazide dose, quantified as the percent change from pre-intake ("OFF" state) to full "ON" state of the Part 3 score of the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

SECONDARY OUTCOMES:
time latency to full "ON" state | Same day of study visit
  Temporal period between L-dopa ingestion and full "ON" state during a single L-dopa challenge test
Part 4 score of the MDS-UPDRS | Same day of study visit
  Motor fluctuations and L-dopa-induced dyskinesia
Maximum observed plasma concentration of L-dopa (Cmax) | Same day of study visit
  The investigators will determine maximum observed plasma concentration (Cmax) directly from serial samples.
Time to maximum observed plasma concentration (Tmax) | Same day of study visit
  The investigators will determine time to maximum observed plasma concentration (Tmax) directly from serial samples.
Area under the L-dopa concentration-time curve (0-3 hours; AUC0-3 h) | Same day as study visit
  The investigators will determine the area under the L-dopa plasma concentration-time curve (0-3 hours; AUC0-3 h).

IPD SHARING:
Plan to Share IPD: Undecided